CLINICAL TRIAL: NCT06599320
Title: Variables for Long-term Success in Implant Dentistry: A Retrospective Cross-sectional Study With a 25 Year Follow-up or More
Brief Title: Variables for Long-term Success in Implant Dentistry
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02279; ITI n 1574_2021 (Other Grant/Funding Number: International Team for Implantology)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dental Implant Failure
Keywords: dental implant; complications
MeSH Terms: interventions — Rehabilitation; Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Partial edentulous patients rehabilitated with at least one dental implant: Partial edentulous patients rehabilitated with at least one dental implant in function for at least 20-years
  Interventions: Other: Oral rehabilitation with dental implants

INTERVENTIONS:
Other: Oral rehabilitation with dental implants — Patients rehabilitated with implant-supported fixed partial dental prostheses

SUMMARY:
The aims of the present retrospective 25-year study of a sample of 459 patients with 753 sandblasted and acid-etched (SLA) titanium oral implants are:

* to assess the clinical parameters at SLA implants after 25 years in function
* to assess the crestal bone levels at SLA implants after 25 years in function
* to assess and compare the microbiological conditions at SLA implants and their adjacent teeth after 25 years of function
* to assess the periodontal conditions in patients having received SLA implants 25 years ago
* to establish a baseline data set for future prospective studies on patients having received SLA implants 25 years ago
* to assess the incidence rates of biological, technical, traumatic failures / complications with SLA implants
* to assess the incidence rates of technical failures / complications with prosthetic components on SLA implants
* to assess the incidence rates of biological, technical, mechanical, esthetic failures / complications with prosthetic reconstructions on SLA implants
* to find potential risk factors for biological failures / complications with SLA implants; i.e. patients having lost their teeth due to different reasons (e.g. partial anodontia, caries, periodontitis, endodontic failure, trauma, vertical root fracture), (ii) to calculate the success rates using different thresholds set as success criteria, (iii) to evaluate the influence of medical conditions and tobacco smoking on the long-term prognosis of titanium oral implants, and (iv) to assess the frequency and quality of maintenance
* to find potential risk factors for mechanical, technical, esthetic failures/complications with reconstructions seated on SLA implants
* to assess the treatment need and utility of implant therapy after 25 years in patients having received SLA implants

DETAILED DESCRIPTION:
Specific aims

The aims of the present retrospective 25-year study of a sample of 459 patients with 753 sandblasted and acid-etched (SLA) titanium oral implants are:

* to assess the clinical parameters at SLA implants after 25 years in function
* to assess the crestal bone levels at SLA implants after 25 years in function
* to assess and compare the microbiological conditions at SLA implants and their adjacent teeth after 25 years of function
* to assess the periodontal conditions in patients having received SLA implants 25 years ago
* to establish a baseline data set for future prospective studies on patients having received SLA implants 25 years ago
* to assess the incidence rates of biological, technical, traumatic failures / complications with SLA implants
* to assess the incidence rates of technical failures / complications with prosthetic components on SLA implants
* to assess the incidence rates of biological, technical, mechanical, esthetic failures / complications with prosthetic reconstructions on SLA implants
* to find potential risk factors for biological failures / complications with SLA implants; i.e. patients having lost their teeth due to different reasons (e.g. partial anodontia, caries, periodontitis, endodontic failure, trauma, vertical root fracture), (ii) to calculate the success rates using different thresholds set as success criteria, (iii) to evaluate the influence of medical conditions and tobacco smoking on the long-term prognosis of titanium oral implants, and (iv) to assess the frequency and quality of maintenance
* to find potential risk factors for mechanical, technical, esthetic failures/complications with reconstructions seated on SLA implants
* to assess the treatment need and utility of implant therapy after 25 years in patients having received SLA implants

Material and methods Out of the pool of patients from the Departments of Oral Surgery and Periodontology and Fixed Prosthodontics at the University of Bern, Switzerland, all patients having received at least one dental implant will be recruited for a comprehensive evaluation 25 years after implant installation and delivery of the reconstruction. The patients had been treated according to a comprehensive treatment strategy prior to the installation of implants and incorporation of reconstructions. All patients were offered maintenance care that was provided either in the School of Dental Medicine, University of Bern, Switzerland, or in the dental practices of the referring dentists at intervals between 3 and 6 months.

All the implants installed were solid screws (SS) with a diameter of 3.3, 4.1 or 4.8 mm, a length between 6-14 mm and a sandblasted and acid-etched surface (SLA) (Straumann® Dental Implant System, Institute Straumann AG, Basel, Switzerland). The implants were placed according to the manufacturer's instructions. The reconstructions were either cemented or screw-retained and consisted of single-unit crowns (SCs) or short-span fixed dental prostheses (FDPs) with or without cantilever extension(s).

ELIGIBILITY:
Inclusion Criteria:

All patients rehabilitated with oral dental implants supporting fixed partial dental prostheses and followed up for at least 20-years.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Out of the pool of patients from the Departments of Oral Surgery and Periodontology and Fixed Prosthodontics at the University of Bern, Switzerland, all patients having received at least one dental implant will be recruited for a comprehensive evaluation 25 years after implant installation and delivery of the reconstruction. The patients had been treated according to a comprehensive treatment strategy prior to the installation of implants and incorporation of reconstructions. All patients were offered maintenance care that was provided either in the School of Dental Medicine, University of Bern, Switzerland, or in the dental practices of the referring dentists at intervals between 3 and 6 months.
  All the implants installed were solid screws (SS) with a diameter of 3.3, 4.1 or 4.8 mm, a length between 6-14 mm and a sandblasted and acid-etched surface (SLA) (Straumann® Dental Implant System, Institute Straumann AG, Basel, Switzerland).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Implant survival rate | 25 years
  percentage of implants in-situ

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schimmel, Study Chair — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buser D, Janner SF, Wittneben JG, Bragger U, Ramseier CA, Salvi GE. 10-year survival and success rates of 511 titanium implants with a sandblasted and acid-etched surface: a retrospective study in 303 partially edentulous patients. Clin Implant Dent Relat Res. 2012 Dec;14(6):839-51. doi: 10.1111/j.1708-8208.2012.00456.x. PMID 22897683